CLINICAL TRIAL: NCT06613087
Title: Effect of Foot Bath on the Severity of Pain, Fatigue and Insomnia in Patients With Acute Renal Failure
Acronym: Foot Bath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Naz Fısgın, Director, Amasya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Naz-682
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Renal Failure; Pain
Keywords: foot bath; insomnia; fatigue
MeSH Terms: conditions — Renal Insufficiency; Pain; Sleep Initiation and Maintenance Disorders; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot bath (Experimental): In the foot bath application, the feet will be kept in water at a constant temperature of 38-40 °C for about 20 minutes. During this time, the water temperature will be checked with a thermometer at intervals. Foot bath applications will be performed for 3 days, on the 2nd, 3rd and 4th days of hospitalization.
  Interventions: Other: Foot bath
- Control (No Intervention): The control group will receive standard care. No intervention will be applied to these patients during the follow-up period, only data collection forms will be applied. Data collection forms will be collected in the same time period as the intervention group.

INTERVENTIONS:
Other: Foot bath — In the foot bath application, the feet will be kept in water at a constant temperature of 38-40 °C for about 20 minutes. During this time, the water temperature will be checked with a thermometer at intervals. Foot bath applications will be performed for 3 days, on the 2nd, 3rd and 4th days of hospitalization.
  Arms: Foot bath

SUMMARY:
One of the non-pharmacological methods that is easily applied, tolerated by the patient, and has no significant side effects is the foot bath. The aim of this study is to determine the effect of a foot bath applied to patients with acute renal failure on the severity of pain, fatigue, and insomnia.

DETAILED DESCRIPTION:
Introduction: One of the non-pharmacological methods that is easily applied, tolerated by the patient, and has no significant side effects is the foot bath.

Objective: The aim of this study is to determine the effect of a foot bath applied to patients with acute renal failure on the severity of pain, fatigue, and insomnia.

Method: The sample of this study will consist of 54 individuals who meet the inclusion criteria among patients with acute renal failure hospitalized in the internal medicine department of a training and research hospital in Amasya. The research data will be collected using a personal information form, numerical pain scale, fatigue severity scale, and insomnia severity index.

Conclusion: In diseases such as acute renal failure that develop suddenly and require hospitalization, it is important to use and evaluate the effectiveness of simple, applicable non-pharmacological methods in order to quickly control the symptoms of patients and ensure their comfort. The study results will contribute to the literature in this field.

ELIGIBILITY:
Inclusion Criteria:

* Those over the age of 18
* Those hospitalized in the internal medicine clinic with a diagnosis of acute renal failure
* Those who speak and understand Turkish
* Those who consent to participate in the study

Exclusion Criteria:

* Those with cognitive dysfunction
* Those diagnosed with chronic renal failure
* Those with wounds on their feet
* Those whose vital signs are not within normal limits (fever, high blood pressure, bradycardia, tachycardia, etc.)
* Those receiving hemodialysis treatment for acute renal failure
* Those taking medication for insomnia
* Those who did not consent to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale | 5 day
  The numerical pain scale was developed to assess the severity of pain. In this scale, the severity of the patient's pain is described with numerical values. Using numerical scales, pain severity is assessed by starting with "0" and grading up to "10". "0" indicates no pain, and "10" indicates unbearable pain. For the scale, the patient is asked to express the level of pain they feel at that moment with a number. The number expressed by the patient is accepted as the severity of the pain felt at that moment.
Fatigue Severity Scale | 5 day
  Fatigue Severity Scale (FSS): FSS is a scale consisting of nine items that evaluate the general effect of fatigue on daily activities. In the scale, individuals are asked to rate the fatigue they have felt throughout the past week from 1 to 7. Each section is scored between 1 (I completely disagree) and 7 (I completely agree). The total score is calculated by taking the average of the nine items. The cut-off value for pathological fatigue is determined as 4 and above. The lower the total score, the less fatigue there is.
Insomnia Severity Index | 5 day
  Insomnia Severity Index: Developed to determine the degree of insomnia symptoms, this can be used in the clinical evaluation of insomnia. It is a five-point Likert-type scale consisting of seven items. Each item is scored between 0 and 4, and the total score varies between 0-28. A score between 0-7 on the scale indicates clinically insignificant insomnia, 8-14 indicates the lower threshold of insomnia, 15-21 indicates clinical insomnia (moderate severity), and 22-28 indicates clinical insomnia (severe).

CONTACTS AND LOCATIONS:
Locations (1):
- AmasyaU, Amasya, Turkey (Türkiye)